CLINICAL TRIAL: NCT04188756
Title: RV Systolic and Diastolic Function and Contractile Reserve Under Acute Exercise and in Response to Chronic Exercise-based Rehabilitation
Acronym: Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniGiessenReserve
Record Dates: First submitted 2019-11-26; First posted 2019-12-06 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Hypertension; Right Heart Failure; Heart Failure; Contractility; RV-arterial Coupling
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients will randomized for exercice (1:1). After 15 weeks the group without exercise will be offered to take part in an exercise training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Other): Group under exercise training for 15 weeks with High intenstiy interval training under medical control
  Interventions: Other: Exercise
- Control (No Intervention): Group with standard care according to current guidelines

INTERVENTIONS:
Other: Exercise — High intensity interval training (rehabilitation) over 15 weeks. Patients will be guided by physicians for exercise training in Pulmonary hypertension
  Arms: Exercise

SUMMARY:
Exercise training in Pulmonary arterial hypertension in the setting of rehabilitation leads to an enormous improvement of functional state and haemodynamics. However the underlying mechanism is still unkown. It is assumed to be relied on Right ventricular contractile reserve, but this has never been proven with goldstandard PV-loop assessment.

Our aim is to evaluate the mechanism leading to the increase in functional state and to evaluate the impact of exercise (acute and chronic) on right ventricular performance

DETAILED DESCRIPTION:
The ability of the RV to increase Ees under exercise is barely understood, and it is not known whether this is accompanied by changes in Eed. Exercise-based rehabilitation programs in PAH patients showed a marked increase in 6 Minute Walk distance and CI; the improvement was, partially higher than the improvement upon targeted PAH medication Several mechanisms may underlie such improvement, in particular a decrease in PVR, improved peripheral muscular function and improved systolic and/or diastolic RV function. To assess the latter aspect in a load-independent fashion, the investigators will perform acute exercising and exercise-based rehabilitation in PAH patients with performance of RV PV loop measurements, which has never been undertaken under this aspect in PAH patients.

Acute exercising: As "physiological response" to acute exercising, an increase in RV Ees is to be expected. However, based on clinical experience and on the surprising finding of an Ees decrease upon volume challenge in patients with low Ees/Ea values, the investigators hypothesize that orientation and extent of the Ees response to acute exercise will depend on the baseline Ees/Ea: patients with well-maintained Ees/Ea values may reveal an increase of Ees in response to acute exercise, whereas patients with RV-PA uncoupling (baseline Ees/Ea < 0.8) may show an acute heterometric adaptation with increase in volumes and decrease in Ees (negative ∆ Ees). Moreover, this study may again provide a novel "threshold of uncoupling" (Ees/Ea ratio), at which the RV response to acute exercising switches from increased to decreased contractility. The investigators will use incremental exercise tests (step or ramp protocol; handgrip protocol) with repeated hemodynamic measurements with right heart catheterization (RHC) and PV-loop catheter. The modified single beat method will be used to calculate Ees and Ea as well as Eed under exercise: the intercept on the x-axis will be predefined by Valsalva maneuver and preload reduction, and this point will be the reference for PV-loop-derived ESPVR to calculate Ees as decribed before. The study will include 42 PAH patients, who will subsequently be entered into the rehabilitation program (for power calculation see below). Similar to the volume challenge study, the hypothesis is that extent and orientation of ∆ Ees upon acute exercise are correlated with baseline Ees/Ea. Primary endpoint: ∆ Ees between baseline and maximum exercise. Secondary endpoints: time to recovery of Ees and RV-EDV after acute exercising, changes in PVR, mPAP, CI, Eed, Ea, Stroke Work, EDP, ESV, EDV and SV. Statistics: the primary endpoint will be analyzed by descriptive statistics, graphical representations with scatterplots, quantitative measures of dependence (Pearson's r or Spearman´s rho) and description of conditional distributions will be used.

Exercise-based rehabilitation - the RESERVE study: The investigators aim to conduct a single center, interventional, randomized, non-blinded, prospective study to evaluate the impact of exercise training on RV-PA- coupling. Every patient will undergo acute exercise testing during first catheterization as described above. Thereafter, patients will be randomly assigned to a control and a training group for chronic exercise in a rehabilitation program. Medication will remain unchanged during the study period. After 15 weeks, RHC and PV-loop assessment at baseline and in response to acute exercise will be repeated. During the study, patients of the control group will not receive any advice on exercise training. Rehabilitation-exercise training will consist of High Intensity Interval Training (HIIT) as described before . Retesting (baseline, response to exercise) will be performed after 15 weeks. Different examinations will be performed at the different visits. Primary endpoint will be the change in baseline Ees over the 15 weeks observation period. Secondary endpoints include the Ees response to acute exercising as well as further PV-loop, cMRI, Echo-derived and functional parameters as detailed in Table 2. Statistics: Continuous variables will be compared using repeated-measures ANOVA for differences between values at baseline and after acute and chronic exercise challenge. The comparisons of characteristics at baseline and after exercise between the two groups, as well as the comparisons of the absolute changes of variables from baseline to post-exercise between groups will be analyzed by adequate descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Consent form,
* men and women> 18 years <75 years
* invasively confirmed chronic PH who have received complete diagnostic evaluation by specialized physicians according to at a center for pulmonary hypertension and were adjusted for 2 months under intensive medical therapy and are stable

Exclusion Criteria:

* Pregnancy or lactation,
* Change in medication during the last 2 months,
* Patients with signs of right heart decompensation, severe walking disturbance,
* No previous invasively confirmation of PH, acute diseases, Infections, fever,
* active myocarditis, unstable angina pectoris, exercise-induced ventricular -arrhythmias, congestive heart failure, significant heart disease, pacemakers, and -hypertrophic obstructive cardiomyopathy, or a highly reduced left ventricular function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint will be the change in baseline Ees over the 15 weeks observation period | over 15 weeks
  Ees(endsystolic elastance) is a measure of coontractility

SECONDARY OUTCOMES:
Global longitudinal strain | over 15 weeks
  Cardiac MRI measures of function, expressed in %
PVR | April 2020 until July 2022
  Right Heart catheter measures of afterload, expressed in Wood Units
Walking distance in 6MW | over 15 weeks
  functional state, expressed in meter
TAPSE, | over 15 weeks
  Echocardiography measure of function, expressed in mm
mPAP | over 15 weeks
  Pressure in Right heart catheter, expressed in mmHg
Cardiac Output | over 15 weeks
  Functional parameter, expressed in liter per minute
T1 mapping | over 15 weeks
  Cardiac MRI parameter, expressed in ms
Fractional area change | over 15 weeks
  Echocardiography measure of function, expressed in %

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Giessen, Giessen, Germany

IPD SHARING:
Plan to Share IPD: No